CLINICAL TRIAL: NCT00567086
Title: A Double-Blind, Placebo-Controlled, Parallel Group Multicenter Study to Assess the Safety, Tolerance and Efficacy of a Single Subcutaneous Dose of TEZAMPANEL in Patients With Acute Migraine
Brief Title: Study to Assess the Safety, Tolerance and Efficacy of Tezampanel in Patients With Acute Migraine
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: TorreyPines Therapeutics (Industry)
Responsible Party: Susan Mellberg, TorreyPines Therapeutics
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NGX424MIG2001
Record Dates: First submitted 2007-12-03; First posted 2007-12-04 (Estimated); Last update posted 2007-12-04 (Estimated); Status verified 2007-12

CONDITIONS: Migraine
Keywords: Migraine
MeSH Terms: conditions — Migraine Disorders | interventions — tezampanel

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- A (Placebo Comparator)
  Interventions: Drug: TEZAMPANEL
- B (Experimental)
  Interventions: Drug: TEZAMPANEL
- C (Experimental)
  Interventions: Drug: TEZAMPANEL
- D (Experimental)
  Interventions: Drug: TEZAMPANEL

INTERVENTIONS:
Drug: TEZAMPANEL — Single Administration of: TEZAMPANEL 40 mg; TEZAMPANEL 70 mg; TEZAMPANEL 100 mg; Placebo (Sterile Water for Injection)
  Other Names: NGX424MIG2001

SUMMARY:
To evaluate the effects of a single sc administration of TEZAMPANEL at one of three different dosage levels compared to placebo, employing traditional measures of efficacy and safety in the treatment of a single episode of acute migraine.

DETAILED DESCRIPTION:
Primary:

• Headache relief (headache response) defined as the percentage of patients in each treatment group who experience a decrease in pain from moderate or severe intensity pre-dose (baseline) to mild or no pain 2 hours after study drug administration and prior to use of rescue medication.

Secondary:

* Percentage of patients in each treatment group who are pain-free two hours after study drug administration, prior to the use of any rescue medication
* Sustained headache response rate (percentage of patients in each treatment group with headache response at Hour 2 and no rescue medication or headache recurrence from 2 through 24 hours)
* Sustained pain-free rate (percentage of patients in each treatment group who are pain free at Hour 2 with no rescue medication or headache recurrence from 2 through 48 hours)
* Recurrence rate (percentage of patients in each treatment group with an Hour 2 mild response or pain-free response who subsequently develop a headache rated as moderate to severe in intensity within 2 to 24 hours)
* Relapse rate (percentage of patients in each treatment group with an Hour 2 pain free response who subsequently develop a headache rated as moderate to severe in intensity within 2 to 48 hours

ELIGIBILITY:
Inclusion Criteria:

* Patients who meet all of the following inclusion criteria at screening should be considered for admission to the study:

  1. Males and females aged 18 to 65 years, inclusive.

     a. Females of childbearing potential must not be at risk for pregnancy during the study.
  2. Patients must meet IHS diagnostic criteria for migraine, with or without aura.
  3. Patients should have a history of 1 to 6 acute migraine headache attacks per month and 1 migraine headache within the past 30 days.
  4. Patients should have at least a 1-year history of migraine headaches.
  5. Patients should have been ≤ 50 years of age at initial migraine onset.
  6. Patients must be able to distinguish migraine headaches as discreet headaches from other headaches, such as tension-type headaches. Additionally, patients should experience at least 48 hours of freedom from headaches between migraine attacks.
  7. Patients must have a complete medical history (including headache history), ECG, and a PE at screening including formal assessments of visual acuity (Snellen chart) and visual field integrity visit.
  8. Patients must be able to comprehend and satisfactorily comply with the protocol requirements, in the opinion of the investigator.

Exclusion Criteria:

* Patients who meet any of the following exclusion criteria at screening will not be eligible for participation in the study.

  1. Patients who also suffer from concomitant frequent, non-migraine headaches ≥6 days/month or who suffer frequent migraine as defined by an average of >6 attacks per month.
  2. Patients who fail to present with a migraine attack for treatment within 30 days of screening.
  3. Patients who have menstrual migraines: migraine attacks occur from days -2 through +3 (Day 1 is the first day of menstruation) of the menses but do not occur the rest of the month.
  4. Patients who have clinically significant active or unstable systemic, renal, hepatic, gastrointestinal, neurological, endocrine, metabolic, or psychiatric disease as determined by medical history and physical examination. Patients who are breast-feeding are excluded. Patients with a history of cardiovascular illness, such as ischemic stroke, ischemic heart disease, Prinzmetal's angina, and hypertension are excluded.
  5. Patients who have received any experimental drugs within one month prior to and one month subsequent to screening.
  6. Patients who have taken a MAOI within 14 days prior to randomization
  7. Patients who are allergic or have shown hypersensitivity to compounds with similar pharmacology to TEZAMPANEL.
  8. Patients who have met the DSM-IV-TR criteria for any significant psychoactive substance use disorder (abuse, dependence, and/or withdrawal) within the past 90 days.
  9. Patients who have a clinically significant abnormal laboratory test result at screening.
  10. Patients who have a clinically notable vital sign abnormality at screening.
  11. Patients will be excluded if 2 consecutive urine drug screenings are positive.
  12. Patients will be excluded if there is evidence of a visual field disturbance.
  13. Patients who have participated in a previous TEZAMPANEL (NGX424 or LY293558) study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 306 (Actual)
Dates: Start 2006-10; Study Completion 2007-08 (Actual)

PRIMARY OUTCOMES:
Headache pain intensity, associated symptoms, functional response questionnaires, time to meaningful pain relief. | 4 Hours

CONTACTS AND LOCATIONS:
Overall Officials: Michael F. Murphy, M.D., Ph.D., Study Chair — TorreyPines Therapeutics
Locations (1):
- National Headache Centers, San Francisco, California, United States